CLINICAL TRIAL: NCT04170504
Title: Efficacy of Chinese Herbal Medicine Qing Re Huo Xue in Patients With Rheumatoid Arthritis: A Randomized Controlled Trial
Brief Title: Efficacy of Chinese Herbal Medicine Qing Re Huo Xue in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018YFC1705203
Record Dates: First submitted 2019-11-14; First posted 2019-11-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Qing Re Huo Xue; Methotrexate; Randomized controlled trial
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qing Re Huo Xue (QRHX) granule plus methotrexate (MTX) (Experimental): QRHX granule 10g bid and methotrexate (MTX) 10 mg once a week for 24 weeks
  Interventions: Drug: Qing Re Huo Xue (QRHX) granule; Drug: Methotrexate
- Qing Re Huo Xue (QRHX) granule placebo plus Methotrexate (MTX) (Placebo Comparator): QRHX granule placebo 10g bid plus Methotrexate (MTX) 10mg once a week for 24 weeks
  Interventions: Drug: Methotrexate; Drug: Qing Re Huo Xue (QRHX) granule placebo

INTERVENTIONS:
Drug: Qing Re Huo Xue (QRHX) granule — Qing Re Huo Xue (QRHX) granule 10g bid for 24 weeks
  Arms: Qing Re Huo Xue (QRHX) granule plus methotrexate (MTX)
Drug: Methotrexate — Oral methotrexate 10 mg per week for 24 weeks.
  Other Names: XINYI Pharm
Drug: Qing Re Huo Xue (QRHX) granule placebo — Qing Re Huo Xue (QRHX) granule placebo 10g bid for 24 weeks
  Arms: Qing Re Huo Xue (QRHX) granule placebo plus Methotrexate (MTX)

SUMMARY:
This study is a multicenter, randomized, double-blinded, placebo-controlled trial with two parallel arms. The aim of the study is to evaluate whether Chinese herbal medicine Qing Re Huo Xue (QRHX) combined with methotrexate (MTX) might be better than Qing Re Huo Xue placebo combined with MTX for patients with active rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
To compare the efficacy and safety of Chinese herbal medicine Qing Re Huo Xue (QRHX) and methotrexate (MTX) for patients with active rheumatoid arthritis (RA), a multicenter, randomized controlled trial will be conducted. Two hundred and four patients with active RA will be randomly allocated (1:1) to treatment with QRHX 10g bid and MTX 10mg once a week for 24 weeks, or MTX plus QRHX placebo. The primary outcome is the bone marrow edema score in Outcome Measures in Rheumatology Clinical Trials RA MRI Scoring (OMERACT-RAMRIS) at week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has had a confirmed diagnosis of rheumatoid arthritis according to 2010 ACR/EULAR RA classification criteria.
2. Subject has a DAS28 CRP disease activity score of >3.2 at screening.
3. Subject also experienced the following signs and symptoms: swelling, joint pain, and heat in the joints.
4. Subject has had no prior exposure to oral glucocorticoids at a daily dose greater than 10 mg or to any biologic agents.
5. Subject may has had previous exposure to nonsteroidal anti-inflammatory drugs (NSAIDs) prior to screening and must be on stable dose.

Exclusion Criteria:

1. History or presence of a clinically significant medical disorder other than RA that, in the opinion of the investigator and medical monitor, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
2. Subject has inflammatory, rheumatological disorders other than RA, where arthritis may be a prominent feature.
3. Subject has received treatment with the prohibited therapies listed in the protocol, or changes to those treatments, within the prescribed timeframe.
4. Pregnant or nursing an infant or with a life partner who is pregnant, nursing, or planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Change in bone marrow edema score from baseline at week 24 in OMERACT RAMRIS | week 0, week 24
  Bone marrow edema score will be assessed by OMERACT-RAMRIS scoring system; minimum value: 0, maximum value: 75; higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in bone erosion score from baseline at week 24 in OMERACT RAMRIS | week 0, week 24
  Bone erosion score will be assessed by OMERACT-RAMRIS scoring system; minimum value: 0, maximum value: 250; higher scores mean a worse outcome.
The proportion of participants with no progression in bone marrow edema and bone erosion | week 24
  No progression in bone marrow edema and bone erosion at week 24 is defined as change in RAMRIS osteitis/erosion score ≤0.
The proportion of participants achieving ACR response (ACR20, ACR50, ACR70) | week 4, week 12, week 24
  The proportion of participants achieving ACR response (ACR20, ACR50, ACR70)
Change in the 28-joint Disease Activity Score in erythrocyte sedimentation rate | week 0, week 4, week 12, week 24
  The improvement of DAS28-ESR and proportion of subjects achieving remission was completed. The subjects achieving remission will be defined as DAS28-ESR &amp;lt;2.6.
Change in Clinical Disease Activity Index (CDAI) | week0, week4, week 12, week 24
  The improvement of CDAI and proportion of subjects achieving remission was completed. The subjects achieving remission will be defined as CDAI <2.8.
Change in Chinese patient-reported activity index with rheumatoid arthritis (CPRI-RA) | week0, week 4, week 12, week 24
  CPRI-RA,The self-rating scale consists of 11 items,Each item was rated 0, 1, 2 and 3 on the scale of asymptomatic to aggravating symptoms, respectively.
Change in Health Assessment Questionnaire Disability Index (HAQ-DI) | week0, week4, week 12, week 24
  The self-rating scale consists of 20 items,Each item was rated 0, 1, 2 and 3 on the scale of asymptomatic to aggravating symptoms, respectively. (range: 0 [best] to 3 [worst])

CONTACTS AND LOCATIONS:
Overall Officials: Quan Jiang, M.D, Principal Investigator — Guang' anmen hospital
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China